CLINICAL TRIAL: NCT00278161
Title: Phase II Study of High Dose Cyclophosphamide and Rituximab in Low Grade and Mantle Cell Lymphoma
Brief Title: Rituximab, Cyclophosphamide, and Pegfilgrastim in Treating Patients With Leukemia or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0260; P50CA096888 (NIH); P30CA006973 (NIH); NA_00041511 (Other: JHMIRB)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Lymphoma
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; B-cell chronic lymphocytic leukemia; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; Waldenstrom macroglobulinemia; prolymphocytic leukemia; stage I marginal zone lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; stage IV marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Leukemia, Prolymphocytic | interventions — pegfilgrastim; Rituximab; Cyclophosphamide

ARMS (1):
- R-HiCy (Experimental): Rituximab (R) and high-dose cyclophosphamide (HiCy) with pegfilgrastim support.
  Interventions: Biological: Pegfilgrastim; Biological: Rituximab; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Pegfilgrastim — 6 mg SQ 24-48 hours after last dose of cyclophosphamide.
  Other Names: Neulasta
Biological: Rituximab — 375 mg/m^2/day on Days 1, 4, 8, 11, 45, and 52.
  Other Names: Rituxan
Drug: Cyclophosphamide — 50 mg/kg/day on Days 15, 16, 17, and 18.
  Other Names: Cytoxan; Cy; CTX

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving rituximab and cyclophosphamide together with pegfilgrastim may be effective in treating leukemia or non-Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well giving rituximab and cyclophosphamide together with pegfilgrastim works in treating patients with B-cell leukemia, low-grade non-Hodgkin's lymphoma, or mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of high-dose cyclophosphamide, rituximab, and pegfilgrastim in patients with B-cell leukemia or low-grade or mantle cell lymphoma.
* Determine the molecular response rate in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive rituximab IV over 30-60 minutes on days 1, 4, 8,11, 45, and 52, cyclophosphamide IV over 1 hour on days 15-18, and pegfilgrastim subcutaneously on day 19 or 20 in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following B-cell leukemias or lymphomas, as defined by World Health Organization criteria:

  * Chronic lymphocytic leukemia/small lymphocytic lymphoma
  * B-cell prolymphocytic leukemia
  * Lymphoplasmacytic leukemia
  * Marginal zone lymphoma (splenic, extranodal, or nodal)
  * Follicular lymphoma (grade 1 or 2)
  * Mantle cell lymphoma
* No more than minimal (approximately 10%) morphologically identifiable cancer cells on bone marrow biopsy

  * When cancer cells are morphologically difficult to distinguish from normal cells, flow cytometry must show no more than 10% identifiable cancer cells
* Must have received ≤ 12 months of prior cytotoxic therapy, achieving at least a partial response NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 75,000/mm^3
* Serum creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2 mg/dL unless secondary to tumor
* AST or ALT < 2 times upper limit of normal
* Normal (≥ 45%) left ventricular cardiac ejection fraction (determined by echocardiogram or MUGA scan)
* DLCO > 50% predicted
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known sensitivity to E. coli-derived products (e.g. filgrastim [G-CSF], insulin, asparaginase, growth hormone, or recombinant interferon alfa-2b) or any treatment study drugs
* No active infections requiring oral or intravenous antibiotics
* No other second malignancy other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix unless the malignancy was localized and treated or resected with > 90% probability of cure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior anti-CD20 therapy allowed provided patient achieved a partial or complete response
* No concurrent steroids during rituximab administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gladstone DE, Bolanos-Meade J, Huff CA, Zahurak M, Flinn I, Borrello I, Luznik L, Fuchs E, Kasamon Y, Matsui W, Powell J, Levitsky H, Brodsky RA, Ambinder R, Jones RJ, Swinnen LJ. High-dose cyclophosphamide and rituximab without stem cell transplant: a feasibility study for low grade B-cell, transformed and mantle cell lymphomas. Leuk Lymphoma. 2011 Nov;52(11):2076-81. doi: 10.3109/10428194.2011.594191. Epub 2011 Jul 14. PMID 21756035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were screen failures. IRB allowed 3 of those participants to be analyzed along with the 78 who were treated as part of the study. Because the 3 additional participants received the exact same protocol intervention, the total population for analysis purposes is 81.
Period: Overall Study
Arm/Group | R-HiCy
Started | 81
Completed | 70
Not Completed | 11
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Arm/Group | R-HiCy
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17
  Male | 59
  Unknown | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Engraftment
Description: Median days to neutrophil and platelet recovery. Neutrophil recovery is defined as absolute neutrophil count >= 500 cells per microliter; platelet recovery is defined as untransfused platelet count >= 20 * 10^9 cells per liter.
Time Frame: Up to 43 days
Measure: Median (Full Range); unit: days
Arm/Group | R-HiCy
Number analyzed (Participants) | 81
days
  Neutrophil | 15 [11 to 32]
  Platelet | 15 [0 to 43]

2. Primary Outcome: Non-relapse Mortality
Description: Number of participants who died for reasons related to protocol treatment.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-HiCy
Number analyzed (Participants) | 81
Participants | 0

3. Primary Outcome: Event-free Survival
Description: Percentage of participants alive without disease relapse.
Time Frame: 5 years
Population: Participants were split into two populations for this outcome only: mantle-cell lymphoma and other low-grade B-cell tumors.
Measure: Number; unit: percentage of participants
Arm/Group | R-HiCy
Number analyzed (Participants) | 81
percentage of participants
  Mantle-cell lymphoma: number analyzed (Participants) | 39
  Mantle-cell lymphoma | 39
  Other low-grade B-cell tumors: number analyzed (Participants) | 42
  Other low-grade B-cell tumors | 40

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse events were assessed at least weekly through Day 60, then at Day 180 and one year.
Arm/Group | R-HiCy
All-Cause Mortality (participants affected / at risk) | 11/81
Serious Adverse Events (participants affected / at risk) | 15/81
Other Adverse Events (participants affected / at risk) | 64/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-HiCy (N=81)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 6 (6)
Fever (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection (unspecified) (Infections and infestations) | 1 (1)
Lipase elevated (Investigations) | 1 (1)
Pain - wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Secondary malignancy - acute myeloid leukemia (Blood and lymphatic system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-HiCy (N=81)
ALT high (Investigations) | 9 (18)
Anemia (Investigations) | 8 (25)
Anorexia (Gastrointestinal disorders) | 17 (18)
Anxiety (Psychiatric disorders) | 10 (10)
AST high (Investigations) | 7 (12)
Bloating (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 10 (10)
Cough (General disorders) | 10 (10)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 21 (22)
Dizziness (Nervous system disorders) | 11 (11)
Edema (Cardiac disorders) | 5 (5)
Fatigue (General disorders) | 30 (33)
Febrile neutropenia (Infections and infestations) | 10 (10)
Fever (Infections and infestations) | 12 (15)
Headache (General disorders) | 16 (21)
Hemorrhoids (Vascular disorders) | 5 (5)
Hiccups (Gastrointestinal disorders) | 5 (5)
Hyperglycemia (Investigations) | 5 (23)
Hypertension (Cardiac disorders) | 8 (8)
Hyponatremia (Investigations) | 4 (7)
Hypotension (Cardiac disorders) | 13 (14)
Insomnia (General disorders) | 12 (12)
Leukopenia (Investigations) | 27 (57)
Lightheadedness (Nervous system disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 45 (59)
Neuropathy (Nervous system disorders) | 13 (14)
Neutropenia (Investigations) | 32 (45)
Orthostatic hypotension (Cardiac disorders) | 5 (6)
Pain - abdomen (General disorders) | 5 (5)
Pain - back (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain - bone (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain - central catheter site (General disorders) | 6 (6)
Pain - hip (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain - mouth (Skin and subcutaneous tissue disorders) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 22 (26)
Rigors (General disorders) | 6 (6)
Diaphoresis (General disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 7 (8)
Thrombocytopenia (Investigations) | 32 (100)
Urinary frequency (Renal and urinary disorders) | 13 (14)
Vomiting (Gastrointestinal disorders) | 33 (40)
Weight gain (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes